CLINICAL TRIAL: NCT00990431
Title: Ablative Fractional Lasers (CO2 and Er:YAG): A Randomized Controlled Blinded Split-face Trial of the Treatment of Peri-orbital Rhytides
Brief Title: Ablative Fractional Lasers to Treat Peri-orbital Rhytides
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laserklinik Karlsruhe (Other)
Responsible Party: Christian Raulin/Professor Dr., Laserklinik Karlsruhe
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LK_05_2009
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Peri-orbital Rhytides
Keywords: skin aging; laser surgery; fractional photothermolysis; comparative study; Ablative fractional treatment of peri-orbital rhytides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon dioxide laser treatment (Active Comparator)
  Interventions: Procedure: Fractional carbon dioxide laser treatment
- Erbium:YAG laser treatment (Active Comparator)
  Interventions: Procedure: Fractional erbium:YAG laser treatment

INTERVENTIONS:
Procedure: Fractional carbon dioxide laser treatment — The CO2 laser (Fraxel Re:pair, Solta Medical Inc., Hayward, CA) employs disposable tips with a diameter of 7 mm and 15 mm, the smaller being used for the peri-orbital region. The laser beam is delivered through multiple deflective and refractive elements and focused to a spot size of approximately 120 µm in diameter at incidence to the skin to deposit an array of laser beams across the surface. Pulse energy varies from 5 to 70 mJ and density from 5 to 70 %. The pulse duration is 10 msec. In the present study, patients received two passes at 15 mJ (1st pass) and 20 mJ (2nd pass), respectively, with a total density of 20 %.
  Arms: Carbon dioxide laser treatment
Procedure: Fractional erbium:YAG laser treatment — The Er:YAG laser used in this study has a fractional handpiece (MCL 30 Dermablate, Asclepion Laser Technologies GmbH, Jena, Germany). By means of a microlens array the laser beam is divided into 13 x 13 small spots with 250 µm diameter each, spread over an area of 13 x 13 mm. A coverage of 5 % of the skin is achieved with a single pass. The pulse duration is 400 μsec. In this trial, we performed 4 passes (resulting in coverage of 20 % of the treated skin) with a total fluence of 60 J/cm² and pulse stacking (6 stacked pulses) to optimize thermal exposure.
  Arms: Erbium:YAG laser treatment

SUMMARY:
Ablative fractional lasers were introduced for treating facial rhytides in an attempt to achieve results comparable to traditional ablative resurfacing but with fewer side effects. However, there is conflicting evidence on how well this goal has generally been achieved as well as on the comparative value of fractional CO2 and Er:YAG lasers. The present study compares these modalities in a randomized controlled blinded split-face study design:

28 patients were enrolled and completed the entire study. Patients were randomly assigned to receive a single treatment on each side of the peri-orbital region, one with a fractional CO2 and one with a fractional Er:YAG laser. The evaluation included Fitzpatrick wrinkle score, profilometric measurement of wrinkle depth (both before and 3 months after treatment) as well as assessment of side effects and patient satisfaction (1, 3, 6 days and 3 months after treatment).

ELIGIBILITY:
Inclusion Criteria:

* age 40-55
* mild to moderate peri-orbital rhytides

Exclusion Criteria:

* unrealistic expectations
* inability to meet follow-up criteria
* Fitzpatrick skin phototype >III
* coagulation disorders or anti-coagulant treatment
* allergy to lidocaine or tetracaine
* oral isotretinoin within the last 6 months
* any active skin disease within the treatment areas (e. g., cancer, autoimmune disease)
* synthetic implants in the treatment area
* facial cosmetic procedures affecting the treatment area within the last 6 months
* photosensitizing medications (e. g., tetracycline, gold)
* history of keloid formation
* pregnancy

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Objective wrinkle depth | 3 months
Wrinkle severity (according to Fitzpatrick´s wrinkle score) | 3 months

SECONDARY OUTCOMES:
Patient satisfaction | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Syrus Karsai, MD, Principal Investigator — Laserklinik Karlsruhe
Locations (1):
- Laserklinik Karlsruhe, Karlsruhe, Germany